CLINICAL TRIAL: NCT06659172
Title: The Effect of Transcutaneous Vagal Nerve Stimulation on the Processing of Visceral Pain Signals: a High Resolution fMRI Study in Healthy Volunteers
Brief Title: Effects of tVNS on Visceral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NL77976.068.21
Record Dates: First submitted 2024-08-01; First posted 2024-10-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Females; Vagus Nerve Stimulation; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Intervention Model Description: The study design is a randomized controlled fMRI study. Subjects will receive two types of stimulation (i.e. taVNS vs sham) during a single scanning visit. The order of stimulation applied during each visit is randomised. Infusion of capsaicin via a nasoduodenal tube will be used as co-intervention.
Who Masked: Participant
Masking Description: Participant will not know the randomization order before starting the fMRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS (Active Comparator): The vagus nerve will be stimulated electrically by using an MRI-safe electrode. The concha of the right ear will be stimulated.
  Interventions: Device: taVNS
- Sham stimulation (Placebo Comparator): The vagus nerve will be stimulated electrically by using an MRI-safe electrode. The earlobe of the right ear will be stimulated.
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — transauricular vagus nerve stimulation

SUMMARY:
Transcutaneous auricular vagal nerve stimulation (taVNS) has shown promise in reducing chronic abdominal pain, such as in irritable bowel syndrome (IBS). This pain is thought to result from a disruption in gut-brain communication involving the vagus nerve. Using brain imaging, we developed a pain model involving capsaicin (the spicy component in red peppers) to study this interaction. This study aims to explore how taVNS affects this pain model in healthy volunteers.

DETAILED DESCRIPTION:
Abdominal pain is often caused by conditions like irritable bowel syndrome (IBS) and functional dyspepsia (FD), which are chronic and can fluctuate daily. IBS and FD affect about 6% and 10% of the general population, respectively. Many patients visiting gastroenterology clinics suffer from these conditions, and pain is the most challenging symptom to manage. Conventional treatments often don't provide lasting relief, affecting patients' quality of life and causing significant socio-economic impact.

The underlying causes of IBS and FD are not well understood, making it difficult to develop effective treatments. These conditions are considered disorders of the gut-brain interaction, involving communication between the gut and brain via the vagus nerve. The vagus nerve sends sensory information from the gut to the brainstem, particularly the nucleus tractus solitarius (NTS), which then communicates with other brain areas involved in pain perception.

The vagus nerve has a branch that innervates the external ear, making it accessible for non-invasive stimulation. Transcutaneous auricular vagal nerve stimulation (taVNS) has been used experimentally for conditions like migraines and fibromyalgia. A recent trial showed that daily taVNS can reduce abdominal pain in adolescents with functional abdominal pain and IBS. Additionally, studies using advanced brain imaging have shown that taVNS activates the NTS. However, it's unclear if this activation is responsible for the pain-relieving effects of taVNS.

New neuroimaging techniques allow for detailed studies of gut-brain communication and the effects of taVNS. Understanding these mechanisms could help develop taVNS as a safe and effective treatment for abdominal pain.

Preliminary Results:

We developed a human pain model using capsaicin (a component of chili peppers) infused into the duodenum to simulate abdominal pain. This model reliably triggers pain and activates brain regions involved in pain perception, including the NTS. This model is useful for studying treatments like taVNS for visceral pain relief.

Clinical Significance:

taVNS is gaining attention as a treatment for various conditions, but its effects are not yet fully understood. This study aims to explore the neurobiological effects of taVNS on visceral pain using advanced imaging techniques. Establishing these effects is crucial for integrating taVNS into clinical practice.

Vagus Nerve Stimulation (VNS):

VNS was first used in 1988 to treat epilepsy with surgically implanted devices. Recently, non-invasive taVNS methods have been developed, targeting the auricular branch of the vagus nerve in the ear. taVNS is safe, well-tolerated, and user-friendly.

Advanced Imaging:

Using 7 Tesla MRI provides higher resolution imaging than standard 1.5 or 3 Tesla scanners, allowing for detailed brain studies. These scanners are becoming more common and are safe for research. In the Netherlands, several institutions use 7 Tesla scanners for patient research without reported adverse effects.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Of female sex;
* Healthy participants (defined as those without a pre-existing medical comorbidity)
* Age between 18 and 40 years;
* BMI between 18 and 30 kg/m2;
* All subjects should use some form of contraception (for IUDs only Mirena is accepted)
* All subjects should be right-handed.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Presence of metallic prostheses, pacemakers, metal clips on blood vessels, metal parts in the eye, an intrauterine device (with the exception of the Mirena IUD), metal braces, facial tattoos and/or other metal objects;
* History of major head trauma or head/brain surgery;
* History of claustrophobia;
* History of severe or chronic cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, haematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol;
* Use of regular medication, including vitamin and iron supplementation, except oral contraceptives, within 14 days prior to start of the study;
* Pregnancy, lactation, wish to become pregnant;
* High alcohol consumption (>15 alcoholic units consumed per week);
* Using drugs of abuse;
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study (to be decided by the principle investigator), in the 180 days prior to the study;
* Participants unable to provide informed consent
* Participants with any systemic disease or medications that may influence the autonomic nervous system (e.g. beta-agonists or Parkinson's disease)
* Current smokers or current use of nicotine in any other way (including E-cigarettes and patches)
* History of clinical anxiety or depression, or a hospital anxiety or depression score >8
* Participants whom score 8 or more on the HADS-questionnaire at study commencement
* Patient whom have cardiovascular conduction problems
* Patient with cochlear implants
* Not meeting any of the inclusion criteria above
* No given permission to register participation in electronic patient file at MUMC+ and to add records of transnasal gastroduodenoscopy
* No given permission to inform incidental findings to the general practitioner
* Any evidence of structural brain abnormalities examined by anatomical MRI will lead to exclusion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Blood oxygenation level dependent BOLD signal activity in the NTS | During fMRI
  Main Outcome Measure
  The main outcome measure is the difference in Blood Oxygen Level Dependent (BOLD) response between taVNS and sham stimulation. The BOLD response is detected using fMRI, which relies on the different magnetic properties of oxygenated and deoxygenated hemoglobin. When neural tissue is more active, it receives increased blood flow, resulting in a higher percentage of oxygenated hemoglobin and a detectable change in the MRI signal. This change, known as the BOLD response, allows us to identify areas of greater neural activity. The BOLD response is a reliable indicator of brain activation.

SECONDARY OUTCOMES:
fMRI results | During fMRI
  BOLD signal activity in the Cingulate Cortex, Insula, Thalamus, Prefrontal Cortex, Primary, Secondary Somatosensory Cortex, Amygdala, Periaqueductal Grey, and Brainstem
fMRI results | During fMRI
  Baseline Cerebral Blood Flow
fMRI results | During fMRI
  Temporal BOLD signal activity (i.e. change over time) in all brain and the above defined regions.
Subjective pain scores | During fMRI
  VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: D. Keszthelyi, Principal Investigator — Maastricht University
Locations (1):
- Maastricht university, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No